CLINICAL TRIAL: NCT06639542
Title: Sexual Agency of Women Who Have Suffered from Incest(s)
Acronym: ASFI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0050_AFSI; N°IDRCB : 2024-A01594-43 (Other: ANSM)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rape Sexual Assault; Incest; Assault; Violence Against Women; Therapy
Keywords: rape; incest; violence; sexual assault; sexuality; agency; psychomotricity; psychomotor therapy
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Case study, qualitative and exploratory approach with prospective research. This study is aimed at voluntary patients referred by the women center.

* The first meeting will be the presentation of a sexo-psychomotor questionnaire, specifically made for this study. Then, if the participant is willing, the enroll for a psychomotor follow-up of 6 sessions personalized with specific objectives defined for the patient,from the questionnaire.
* These therapy sessions can be renewed in discussion with the woman if we feel they would benefit from further follow-up. The psychomotor sessions last around 45 minutes and take place once every 15 days or 3 weeks with a variety of therapeutical techniques. This interval between sessions allows time for integration of the aspects addressed during the proposals, while ensuring continuity in the follow-up. They are aimed at developing body and emotional awareness, to help patients get to know themselves better, and experience moments in full awareness
* End-of-follow interview with taking the questionnaire a second time, to determine, with the woman, any benefits of the "sex-psychomotor" care. The women will be supported in completing the questionnaire again, as they were during the initial session.

DETAILED DESCRIPTION:
First meeting with the presentation of a "sexo-psychomotor" questionnaire targeting patients' sexual agency. This questionnaire was made specifically for this study, based on the levels of sexual agency established by Denise Medico and Julie Lavigne.

7 Levels of sexual agency are described, with associated levels 4 and 5 (detailed and explained in the CRF document):

* Level 1 : Corporeality and self-presence. We'll be dealing with the participants' bodily sensations (sensory, tonic, etc.): exploring them, identifying them, naming them, and becoming aware of any associated thoughts and representations. The aim would be to validate and develop their physical and emotional awareness, identify what they do or don't want, and enable them to explore how to welcome their feelings.
* Level 2 : Sexual subjectivity. We will be working on the participants' self-definition regarding their gender and associated representations, their sexual and romantic orientation, and their experiences and feelings about their sexuality (sensations, emotions, representations, fantasies). The aim would be to enrich their body knowledge and representations (body schema and body image), to identify what is negative for them to distance themselves from it/protect themselves from it, and to clarify what is meaningful, positive, and beneficial for them to promote it.
* Level 3 : Affirmation and identity. Based on the activities, situations, or elements identified as positive/pleasant/appreciated by the participants in the previous levels, we seek to give value to their feelings, tastes, and choices, and to support their expression for themselves and others (especially intimate partners).
* Level 4 and 5 : Intimacy and relational and communicational skills. The aim will be to reinforce the interpersonal and communication skills of participants in their intimate time by identifying and expressing their needs as well as their partners. We want to increase their communication and empathy.
* Level 6 : Mutuality and play. We want to develop the playfulness of the participants to boost both the discovery between their partners and them during intimacy (not exclusively)
* Level 7 : Perspective of transcendence. For this last level, after all the work done previously, we want the participant to be spontaneous and independent about their agency.

These different levels build on each other and are rooted in women's physical and emotional experiences. In the questionnaire I suggest, levels 4 and 5 (Intimacy and Relational and Communicative Capacities) are combined for practical reasons, as the notions are particularly intertwined. Some aspects of these different levels may also overlap.

The questionnaire will be used as an initial assessment to determine more specific sex therapy goals based on each woman's sexual agency and to establish whether she wants to address her sexual agency after this assessment.

The different levels of agency in this questionnaire are assessed through different questions (from 2 to 10 questions depending on the level), which participants can answer using numerical scales from 1 to 10. The scales have been constructed in such a way that the lower the agency assessed, the lower the score. These different numerical values can then be added together to obtain an overall score for each level.

For instance, in the first level of sexual agency "Corporeality and self-presence", the highest score of agency will be 50.

However, some questions can't be answered with a numerical scale : The participant will have to color a figure or circle their emotions or answers, that couldn't have been relevant with a numerical scale. Some questions may be intrusive, the participants are free to tick the box "I am not concerned" or "I do not wish to answer". This answer will also be apprehended on a qualitative assessment.

An overall agency score will be determined by incorporating all the questions for which a quantitative assessment is possible, with a proportional coefficient for each level (the number of questions is not the same for each level). This overall score will be out of 60 points (10 points per level).

As it is not possible to score all the responses, I will carry out a qualitative and comparative analysis of the participants' responses for which numerical scoring is not possible.

If the participant is interested: set up a 6-session "sexo-psychomotor" follow-up based on the therapeutic objectives determined via the questionnaire.

The content of the sessions will not necessarily be the same from one patient to the other, as it is unlikely that all the women referred to us will have the same needs. Not all women will come to us with the same "background" and similar demands, which means that we need to adapt the support we offer.

To determine objectives and therapeutic proposals tailored to each patient, we will use the results of the questionnaire according to each theme or level of agency.

If some of the women assessed have a low level of sexual agency in level 1 (physicality and self-presence), we'll work on this axis first. Depending on their progress, we'll stay on this theme or move on to the next.

It should be noted that the limits between the different levels are permeable, the levels can overlap and the therapeutic objectives prepare and enrich the following ones. Finally, certain therapeutic mediations can be used to develop different levels of sexual agency, although the objectives to which they respond evolve in parallel with the participants' acquisition of a higher level of sexual agency.

Thus, the follow-up suggested in this study would have the particularity of moving towards sex-therapeutic objectives with psychomotor care and mediation (described above), hence the name "sex-psychomotricity".

Each session is divided into three parts:

* a first time of exchange (the participant's mood, expression of emotional or physical feelings, remarks in connection with the previous session(s), etc.).
* a second psycho-physical phase, using psychomotor mediation(s) (relaxation...).
* a third and final phase of verbalization/elaboration of what has been experienced during the mind-body session, with a link to the sexo therapy objectives and possible "infusion" into the field of sexuality.

End-of-care interview, with a second round of questionnaires, to determine, in discussion with the woman, any benefits of the "sex-psychomotor" care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Women who have suffered from incest or rape
* Speak and understand French

Exclusion Criteria:

* Refusal to participate
* Non french-speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women receiving care at the Women's center (Maison des femmes) and referred for "sexo psychomotor therapy"
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Demographic information | [1day]
  Age of the participant
Follow up at the Women's center | [1day]
  how long they have been followed up at the center; what kind of therapy or help they are receiving
Type of violence | [1day]
  description of the violence (incest, rape or any other type of violence) the participant went through
Agency questionnaire | [1 day]
  Agency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Maison des femmes, Saint-Denis, Seine Saint Denis, France

IPD SHARING:
Plan to Share IPD: No